CLINICAL TRIAL: NCT05607355
Title: Measurement of Spinal Mobilization Biomechanical Parameters in the Preschool Pediatric Population
Brief Title: Measurement of Spinal Mobilization in Pediatric Population
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Fondation Chiropratique du Québec (Other); Canadian Chiropractic Research Fondation (Unknown)
Responsible Party: Principal Investigator, Isabelle Pagé, Professor, Université du Québec à Trois-Rivières
Other Study IDs: UQTR_PEDS_MOB_2022-2023
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pediatric ALL
Keywords: Manual therapy; Chiropractic; Vertebral mobilisation; Pediatric; Biomechanics; Safety
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cross-sectional study is to measure the biomechanical parameters during a vertebral mobilization delivered by chiropractors on patients of five years old of age and younger. The main questions it aims to answer are:

* What is the force and rate of force application of spinal mobilizations in children consulting in chiropractic?
* What are the adverse events observed by legal tutors immediately following the intervention received by the child?

Participants will receive the clinically indicated spinal mobilization by their treating chiropractor. The chiropractor will have a small sensor on the finger during the delivery of the spinal mobilization. The legal tutor will complete a questionnaire immediately after the intervention to report adverse events.

DETAILED DESCRIPTION:
Scope: Number of parents consulting complementary and alternative medicine practitioners for their children's health is increasing. Spinal mobilization is commonly provided by these practitioners, including chiropractors, to address health disorders in children. Spinal mobilization involves the application of a controlled force to a vertebra using a slow speed and is considered an appropriate technique in young children. Despite the popularity of spinal mobilization in the pediatric population, only a paucity of data exists on its biomechanics. One study has evaluated the force used by chiropractors on manikins and one study calculated theoretical values of the maximum force that should be applied in function of the patient age. To date, no studies have characterized spinal mobilization biomechanics using a pragmatic approach: measurement directly at the clinician's hands during spinal mobilization delivered on real pediatric patients.

Purpose: The aims are to (1) measure the biomechanical parameters during spinal mobilization delivered by chiropractors on patients of 5 years of age or younger and (2) to report immediate adverse events.

Methodology:

Design: This research proposal is a pragmatic cross-sectional study. Participants: Patients seeking care at our collaborating chiropractic clinics and aged between 0 (newborn) and 5 years old will be recruited. Spinal mobilization will have to be clinically indicated. A total of 60 participants will be recruited.

Experiment: To measure spinal mobilization parameters, the chiropractor will wear a small sensor on their finger tip used to deliver the spinal mobilization (MedicalSensor 9811E, Tekscan, Boston, US). The sensor record force by time data using a 100 Hz acquisition frequency. Legal guardians will complete a short online questionnaire (pediatric version of the SafetyNet system) immediately following the intervention to report any adverse events. Participant characteristics (age, weight, height, sex, reason to seek care) will also be collected.

Primary outcomes: Spinal mobilization peak force and rate of force applications (i.e., speed).

Secondary outcomes: Immediate adverse events observed by the legal guardian. Analyses: The sample of participants will be descriptively analyzed. The mean, range and standard deviation of the peak force and rate of force applications measured during the spinal mobilizations will be reported. Adverse events frequency and nature will be reported. Exploratory analyzes will be conducted to explore the associations between participants' characteristics, treated region of the spine and spinal mobilization's peak force and rate of force applications

ELIGIBILITY:
Inclusion criteria :

* Being aged between 0 (newborn) and 5 years old
* Consulting a chiropractor involved in the study
* Having at spinal mobilization included in the care plan.

Exclusion Criteria:

- Not requiring a spinal mobilization on the day of data collection.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 60 children 5 years old and less will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Spinal mobilization force | During the intervention.
  For each spinal mobilization delivered by the chiropractor on the participant, the peak force will be measured.
Spinal mobilization rate of force application | During the intervention.
  For each spinal mobilization delivered by the chiropractor on the participant, the rate of force will be measured.

SECONDARY OUTCOMES:
Adverse events | 5-min following the intervention
  Adverse events of the intervention observed by the legal guardian of the participant will be reported using a validated questionnaire (pediatric verson of the SafetyNet reporting system).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pagé, PhD, Principal Investigator — Département de Chiropratique
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Triano JJ, Lester S, Starmer D, Hewitt EG. Manipulation Peak Forces Across Spinal Regions for Children Using Mannequin Simulators. J Manipulative Physiol Ther. 2017 Mar-Apr;40(3):139-146. doi: 10.1016/j.jmpt.2017.01.001. Epub 2017 Mar 6. PMID 28274487
- [Background] Marchand AM. A Proposed Model With Possible Implications for Safety and Technique Adaptations for Chiropractic Spinal Manipulative Therapy for Infants and Children. J Manipulative Physiol Ther. 2015 Nov-Dec;38(9):713-726. doi: 10.1016/j.jmpt.2013.05.015. Epub 2013 Jul 8. PMID 23845198
- [Background] Pohlman KA, Carroll L, Tsuyuki RT, Hartling L, Vohra S. Comparison of active versus passive surveillance adverse event reporting in a paediatric ambulatory chiropractic care setting: a cluster randomised controlled trial. BMJ Open Qual. 2020 Nov;9(4):e000972. doi: 10.1136/bmjoq-2020-000972. PMID 33203708
- See also: Journal interview about the study — https://neo.uqtr.ca/2022/04/25/lingenierie-pour-optimiser-le-traitement-chiropratique-aupres-des-jeunes-enfants/